CLINICAL TRIAL: NCT05921994
Title: Long Term observAtional, Prospective, Multicenter Study to Collect iN a Real-world populatIon Data on the treatMent Pattern of secukinumAb in Adult Patients With Moderate to Severe Hidradenitis Suppurativa (HS) (ANIMA)
Brief Title: Long Term Observational Study to Collect in a Real-world populatIon Data on the Treatment Pattern of secukinumAb in Adult Patients With Moderate to Severe Hidradenitis Suppurativa.
Acronym: ANIMA
Status: Active, not recruiting | Type: Observational
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Other Study IDs: CAIN457MDE01
Record Dates: First submitted 2023-06-16; First posted 2023-06-28 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Hidradenitis Suppurativa
Keywords: Hidradenitis suppurativa; HS; secukinumab; Germany; NIS
MeSH Terms: conditions — Hidradenitis Suppurativa | interventions — secukinumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- secukinumab: Patients being treated for HS with secukinumab according to the summary of product characteristics (SmPC), after the approval of secukinumab has been granted in this indication.
  Interventions: Other: secukinumab

INTERVENTIONS:
Other: secukinumab — Prospective observational study. There is no treatment allocation. Patients administered secukinumab by prescription and administered according to the SmPC.

SUMMARY:
The purpose of this observational, prospective, non-interventional, multicenter, open-label, single arm study in Hidradenitis suppurativa (HS) is to assess the treatment pattern of secukinumab in a flexible dosing regimen and decision influencing factors for flexible dosing in a real-world population over 2 years.

DETAILED DESCRIPTION:
The study will collect data from patients during routine secukinumab treatment and will be representative of the real-world patient population eligible for secukinumab treatment in Germany.

In order to attain widespread representation of health care practices related to the use of secukinumab in the approved indication of moderate to severe HS, a broad spectrum of dermatology practices and clinics who are treating patients with HS across Germany will be included.

ELIGIBILITY:
Inclusion Criteria:

Patients eligible for inclusion in this study have to fulfill all of the following criteria at enrollment:

1. Patients who provide written informed consent to participate in the study
2. Male and female patients with ≥18 years of age
3. Diagnosis of clinically unequivocal moderate to severe HS
4. Patients for whom a therapy with secukinumab is medically indicated
5. Documented decision for treatment with marketed secukinumab regardless of this noninterventional study
6. Treatment with secukinumab according to the latest version of SmPC
7. Initial treatment with marketed secukinumab planned for up to 1 week before the baseline visit

Exclusion Criteria:

Patients fulfilling any of the following criteria at enrollment are not eligible for inclusion in this study. No additional exclusions may be applied by the investigator, in order to ensure that the study population will be representative of all eligible patients:

1. Patients who have any contraindications, such as a history of or active inflammatory bowel disease (Crohn´s disease, ulcerative colitis), and are not eligible for treatment with secukinumab according to the SmPC
2. Any medical or psychological condition in the treating physician's opinion which may prevent the patient from the study participation
3. Simultaneous participation in any investigational trial or simultaneous participation in another Novartis-sponsored non-interventional study with secukinumab
4. Previous exposure to IL-17 inhibitors
5. For biologic-naïve patients, previous exposure to another biologic drug, such as anti-TNF-α inhibitors

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients, being treated for HS with secukinumab according to the summary of product characteristics (SmPC), after the approval of secukinumab has been granted in this indication.
Sampling Method: Non-Probability Sample
Enrollment: 425 (Actual)
Dates: Start 2023-08-10 (Actual); Primary Completion 2027-03-31 (Estimated); Study Completion 2027-03-31 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients receiving up-titration | Up to 24 months
  Proportion of patients receiving up-titration (q4w-to-q2w)
Proportion of patients receiving down-titration | Up to 24 months
  Proportion of patients receiving down-titration (q2w-to-q4w)
Time to up-titration and down-titration | Up to 2 years
  Time to up-titration and down-titration
Duration of q4w treatment with secukinumab after dose reduction | Up to 2 years
  Duration of q4w treatment with secukinumab after dose reduction
Proportion of patients who receive more than one up-and/or down titration | Up to 24 months
  Proportion of patients who receive more than one up-and/or down titration
Proportion of patients receiving HS-specific concomitant treatments in combination with secukinumab | Up to 2 years
  Proportion of patients receiving HS-specific concomitant treatments in combination with secukinumab
Number and type of surgical interventions | Up to 2 years
  Number and type of surgical interventions
  * minor and major surgical excision;
  * inpatient, outpatient
Proportion of patients achieving 55% reduction in IHS4 (IHS4-55) | Up to 24 months
  The IHS4 is an exclusively physician-based, clinical scoring system for dynamic assessment of HS severity.
  HS severity is calculated based on the number of lesions multiplied by their respective score: the IHS4 score (points) = (number of nodules multiplied by 1) + (number of abscesses multiplied by 2) + [number of draining tunnels (fistulae/sinuses) multiplied by 4]. A score of 3 or less signifies mild HS, a score of 4-10 signifies moderate HS and a score of 11 or higher signifies severe HS
mean change of International Hidradenitis Suppurativa Severity Score System (IHS4) | Up to 24 months
  The IHS4 is an exclusively physician-based, clinical scoring system for dynamic assessment of HS severity.
  HS severity is calculated based on the number of lesions multiplied by their respective score: the IHS4 score (points) = (number of nodules multiplied by 1) + (number of abscesses multiplied by 2) + [number of draining tunnels (fistulae/sinuses) multiplied by 4]. A score of 3 or less signifies mild HS, a score of 4-10 signifies moderate HS and a score of 11 or higher signifies severe HS
Proportion of patients achieving a 5-point reduction of their Dermatology Life Quality Index (DLQI) questionnaire | Up to 24 months
  The DLQI is a 10-item general dermatology disability index designed to assess health-related quality of life (HRQoL) in adult subjects with skin diseases such as eczema, psoriasis, acne, and viral warts. The measure is self-administered and includes domains of daily activities, leisure, personal relationships, symptoms and feelings, treatment, and work/school.
  Each item has four response categories ranging from 0 (not at all) to 3 (very much). "Not relevant" is also a valid response and is scored as 0. The DLQI total score is a sum of the 10 questions. Scores range from 0 to 30, with higher scores indicating greater HRQoL impairment.
Mean reduction of Abscesses and inflammatory nodules (AN) count | Up to 24 months
  Mean reduction of Abscesses and inflammatory nodules (AN) count
Proportion of patients achieving a 30% reduction of pain Numerical Rating scale 30 (NRS30) | Up to 24 months
  The NRS is a segmented numeric version of the visual analog scale (VAS) in which a respondent selects a whole number (0-10 integers) that best reflects the intensity of their pain ranging from 0 (no skin pain) to 10 (skin pain as bad as you can imagine). To assess this, the patient should concentrate on the pain that his/her skin lesions generate. The Patient's Global Assessment of Skin Pain - NRS will be completed by the subject electronically via a web-based application or in paper form.

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (75):
- Germany (75):
  - Novartis Investigative Site, Freiburg im Breisgau, Baden-Wurttemberg
  - Novartis Investigative Site, Rheinstetten, Baden-Wurttemberg
  - Novartis Investigative Site, Kulmbach, Bavaria
  - Novartis Investigative Site, Lauf an der Pegnitz, Bavaria
  - Novartis Investigative Site, Nuremberg, Bavaria
  - Novartis Investigative Site, Hamburg, Hamburg
  - Novartis Investigative Site, Lingen Ems, Lower Saxony
  - Novartis Investigative Site, Kröpelin, Mecklenburg-Vorpommern
  - Novartis Investigative Site, Krefeld, North Rhine-Westphalia
  - Novartis Investigative Site, Mainz, Rhineland-Palatinate
  - Novartis Investigative Site, Dresden, Saxony
  - Novartis Investigative Site, Leipzig, Saxony
  - Novartis Investigative Site, Wittenberg, Saxony-Anhalt
  - Novartis Investigative Site, Aachen
  - Novartis Investigative Site, Ahaus
  - Novartis Investigative Site, Annaberg-Buchholz
  - Novartis Investigative Site, Bad Steben
  - Novartis Investigative Site, Baden-Baden
  - Novartis Investigative Site, Bergen
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Bielefeld
  - Novartis Investigative Site, Bochum
  - Novartis Investigative Site, Bonn
  - Novartis Investigative Site, Brandenburg
  - Novartis Investigative Site, Bremen
  - Novartis Investigative Site, Buxtehude
  - Novartis Investigative Site, Bückeburg
  - Novartis Investigative Site, Chemnitz
  - Novartis Investigative Site, Cologne
  - Novartis Investigative Site, Delitzsch
  - Novartis Investigative Site, Dessau
  - Novartis Investigative Site, Dorsten
  - Novartis Investigative Site, Dortmund
  - Novartis Investigative Site, Dresden
  - Novartis Investigative Site, Düren
  - Novartis Investigative Site, Emsdetten
  - Novartis Investigative Site, Erlangen
  - Novartis Investigative Site, Falkenberg
  - Novartis Investigative Site, Falkensee
  - Novartis Investigative Site, Freising
  - Novartis Investigative Site, Geilenkirchen
  - Novartis Investigative Site, Gera
  - Novartis Investigative Site, Gernsbach
  - Novartis Investigative Site, Gladbeck
  - Novartis Investigative Site, Großenhain
  - Novartis Investigative Site, Hamburg
  - Novartis Investigative Site, Hanover
  - Novartis Investigative Site, Hasfurt
  - Novartis Investigative Site, Haslach im Kinzigtal
  - Novartis Investigative Site, Hofgeismar
  - Novartis Investigative Site, Jena
  - Novartis Investigative Site, Jülich
  - Novartis Investigative Site, Karlsruhe
  - Novartis Investigative Site, Kempen
  - Novartis Investigative Site, Lübeck
  - Novartis Investigative Site, Magdeburg
  - Novartis Investigative Site, Mainz
  - Novartis Investigative Site, Marburg
  - Novartis Investigative Site, Minden
  - Novartis Investigative Site, Mönchengladbach
  - Novartis Investigative Site, Neu Wulmstorf
  - Novartis Investigative Site, Nuremberg
  - Novartis Investigative Site, Oberasbach
  - Novartis Investigative Site, Oelde
  - Novartis Investigative Site, Panketal
  - Novartis Investigative Site, Peitz
  - Novartis Investigative Site, Potsdam
  - Novartis Investigative Site, Remscheid
  - Novartis Investigative Site, Selters
  - Novartis Investigative Site, Simmern
  - Novartis Investigative Site, Soest
  - Novartis Investigative Site, Stolberg
  - Novartis Investigative Site, Unna
  - Novartis Investigative Site, Wittlich
  - Novartis Investigative Site, Wuppertal

IPD SHARING:
Plan to Share IPD: No